CLINICAL TRIAL: NCT02928367
Title: The Effect of Leukocyte Dna mEthylation and micRoBIOME Diversity on Host Defense Mechanisms During Community-acquired Pneumonia
Brief Title: The Effect of Leukocyte Dna mEthylation and micRoBIOME Diversity on Host Defense Mechanisms During Community-acquired Pneumonia (ELDER-BIOME)
Acronym: ELDER-BIOME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, T. van der Poll, prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL57847.018.16
Record Dates: First submitted 2016-10-06; First posted 2016-10-10 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — feces, nasofaryngeal swabs, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pneumonia patients: rectal swab (4x) divided over two time points (day 0 and day 28) nasopharyngeal swab (2x) divided over two time points (day 0 and day 28) blood draw (90ml) divided over two time points (day 0 and day 28)
  Interventions: Other: rectal swab; Other: nasopharyngeal swab; Other: blood draw
- Healthy subjects: rectal swab (2x) nasopharyngeal swab (2x) blood draw (70ml)
  Interventions: Other: rectal swab; Other: nasopharyngeal swab; Other: blood draw

INTERVENTIONS:
Other: rectal swab — rectal swab at baseline visit (2x) and at day 28 (2x) OR rectal swab at single timepoint (2x) (healthy volunteers)
Other: nasopharyngeal swab — nasopharyngeal swab at baseline visit (1x) and at day 28 (1x) OR nasopharyngeal swab at single timepoint (2x) (healthy volunteers)
Other: blood draw — blood draw at baseline visit (45ml) and at day 28 (45ml) (pneumonia patients) OR single blood draw (70ml) (healthy volunteers)

SUMMARY:
Community-acquired pneumonia (CAP) represents a major health care problem and mortality and morbidity associated with severe pneumonia remain considerable, despite state of the art care.

While the role of altered DNA methylation in cancer has been widely studied, knowledge of its impact on antibacterial defense is highly limited. In addition, recent preclinical studies showed that the gut and respiratory microbiota contributes to host defense against bacterial pneumonia.

This study aims to explore a completely novel research area linking the extent of DNA methylation in blood leukocyte (monocytes and neutrophils) and function of gut and respiratory microbiota on the influence of innate immune responses to and host defense against CAP

DETAILED DESCRIPTION:
Rationale:

Community-acquired pneumonia (CAP) represents a major health care problem and mortality and morbidity associated with severe pneumonia remain considerable, despite state of the art care.

While the role of altered DNA methylation in cancer has been widely studied, knowledge of its impact on antibacterial defense is highly limited. In addition, recent preclinical studies showed that the gut and respiratory microbiota contributes to host defense against bacterial pneumonia.

This study aims to explore a completely novel research area linking the extent of DNA methylation in blood leukocyte (monocytes and neutrophils) and function of gut and respiratory microbiota on the influence of innate immune responses to and host defense against CAP.

Primary Objectives:

1. To obtain insight in the role of altered DNA methylation in blood leukocytes (monocytes and neutrophils) in innate immune responses and host defense in patients with CAP.
2. To determine the composition and function of the gut and respiratory microbiota in patients with CAP.

Secondary Objective:

1. To assess the influence of the gut microbiota on leukocyte DNA methylation in patients with CAP

Study design:

Observational study among patients with CAP at the Emergency Department and Internal Medicine Ward of the Academic Medical Center Amsterdam

Study population:

231 CAP patients and 115 healthy subjects above 18 years of age.

Methods:

From above mentioned patients and healthy volunteers, a maximum of 90 ml of blood will be drawn to analyze DNA methylation patterns of purified monocytes and neutrophils, which will be analyzed in connection with DNA methyltransferase and ten eleven translocation (TET) activity, RNA gene expression and a selection of standard innate immune function tests. Moreover, isolated monocytes and neutrophils from admission samples will be stimulated in vitro with Streptococcus pneumoniae and Klebsiella pneumoniae. In addition, rectal and nasopharyngeal swabs will be obtained to investigate the role of the gut and respiratory microbiota composition and function. Patient material will be obtained upon inclusion and on day 28, when patients will be seen in the outpatient clinic for follow up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Participating in this observational study will not benefit the participants and healthy volunteers. The study will provide information about the influence of leukocyte DNA methylation as well as the gut and respiratory microbiota on host defense mechanisms during CAP. The knowledge obtained can potentially benefit CAP patients in the future by providing alternative immune modulating treatment options that modify the host response. The burden and risks for patients participating in the ELDER-BIOME study is minimal. The investigators will take 90ml of blood, 4 rectal swabs and 2 nasopharyngeal swabs divided over two time-points (day of presentation and day 28 post presentation). Healthy volunteers will be subjected to one blood draw (70 ml) and 2 rectal - and 2 nasopharyngeal swabs at one time-point.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of a new episode of acute respiratory tract infection
* Primary reason for presentation is clinical suspicion of a new episode of acute respiratory infection; admission to the hospital is NOT a requirement
* Evident new or progressive infiltrate, consolidation, cavitation, or pleural effusion on the chest X ray or CT scan made for diagnostic (non-research) purposes
* Onset of the following symptoms within the last 7 days:
* At least one respiratory symptom (cough, sore throat, runny or congested nose, dyspnea)
* At least one systemic symptom (fever, headache, muscle ache, sweats or chills or tiredness).

Exclusion Criteria:

* Patient lacks capacity to provide informed consent
* No informed consent is provided by patient
* Patient has been transferred from another hospital
* Patient is enrolled in an interventional clinical study of an anti-infective or immunomodulatory therapy
* Patient has received any type of oral or systemic antibiotics for more than 48 hours prior to hospital presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults presenting at the Academic Medical Center with a suspected new episode of community acquired pneumonia will be screened for eligibility for the ELDER-BIOME study according to the following scheme:
Sampling Method: Probability Sample
Enrollment: 231 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Alterations in leukocyte DNA methylation | day 0

SECONDARY OUTCOMES:
Composition and function of the gut and nasopharyngeal microbiota | day 0
Alterations in leukocyte DNA methylation | day 28
Composition and function of the gut and nasopharyngeal microbiota | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Tom van der Poll, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center - University of Amsterdam, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Brands X, van Engelen TSR, de Vries FMC, Haak BW, Klarenbeek AM, Kanglie MMNP, van den Berk IAH, Schuurman AR, Peters-Sengers H, Otto NA, Faber DR, Lutter R, Scicluna BP, Stoker J, Prins JM, Joost Wiersinga W, van der Poll T. Association of Hyperferritinemia With Distinct Host Response Aberrations in Patients With Community-Acquired Pneumonia. J Infect Dis. 2022 Jun 1;225(11):2023-2032. doi: 10.1093/infdis/jiac013. PMID 35100411
- [Derived] Brands X, Haak BW, Klarenbeek AM, Butler J, Uhel F, Qin W, Otto NA, Jakobs ME, Faber DR, Lutter R, Wiersinga WJ, van der Poll T, Scicluna BP. An epigenetic and transcriptomic signature of immune tolerance in human monocytes through multi-omics integration. Genome Med. 2021 Aug 16;13(1):131. doi: 10.1186/s13073-021-00948-1. PMID 34399830
- [Derived] Brands X, de Vries FMC, Uhel F, Haak BW, Peters-Sengers H, Schuurman AR, van Engelen TSR, Lutter R, Cremer OL, Bonten MJ, Schultz MJ, Scicluna BP, van der Poll T; MARS Consortium. Plasma Ferritin as Marker of Macrophage Activation-Like Syndrome in Critically Ill Patients With Community-Acquired Pneumonia. Crit Care Med. 2021 Nov 1;49(11):1901-1911. doi: 10.1097/CCM.0000000000005072. PMID 33935163